CLINICAL TRIAL: NCT05530798
Title: Contrast Enhanced Ultrasound for The Evaluation of Intraoperative Spinal Cord Injury Following Surgical Decompression of a Chronically Compressed Spinal Cord
Brief Title: CEUS For Intraoperative Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: South Carolina Spinal Cord Injury Research Fund (Unknown)
Responsible Party: Principal Investigator, Stephen Kalhorn, Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00120959
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-11

CONDITIONS: Spine Disease; Spinal Stenosis; Spinal Injury; Spinal Cord Diseases; Spinal Cord Injuries; Spinal Cord Compression; Spine Degeneration
Keywords: Contrast Enhanced Ultrasound; CEUS
MeSH Terms: conditions — Spinal Diseases; Spinal Stenosis; Spinal Injuries; Spinal Cord Diseases; Spinal Cord Injuries; Spinal Cord Compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Contrast Enhanced Ultrasound Arm (Experimental)
  Interventions: Device: Definity Perflutren Lipid Microsphere Ultrasound Contrast

INTERVENTIONS:
Device: Definity Perflutren Lipid Microsphere Ultrasound Contrast — 1. Before the spinal decompression surgery has started, the study team will inject the ultrasound contrast to visualize the spinal cord prior to decompression of the spinal cord.
  2. After the spinal cord has been decompressed, the study team will inject the ultrasound contrast to visualize the spinal cord directly after decompression of the spinal cord.
  3. Prior to completion and closure of the incision, the study team will once more inject the ultrasound contrast to visualize the spinal cord.
  4. A member of the research team will follow up with study participants within a week of the procedure by phone. The research staff will also review the participants' medical record for up to 360 days after your procedure to collect information on clinical outcomes and any additional treatments, tests or procedures the study participants may have had.

SUMMARY:
Spinal cord injury following posterior decompression in patients suffering from chronic, cervicothoracic spinal cord compression is a known complication with multiple etiologies. Currently, intraoperative neuromonitoring (IONM) remains the gold standard for predicting and preventing post-operative deficits from these procedures. However, there is a paucity in the field of spine surgery for further, non-invasive biomarkers that can help detect and prognosticate the degree of spinal cord injury intraoperatively. Contrast enhanced ultrasound (CEUS) is a radiation free imaging modality that utilizes nanobubble technology to allow for visualization of the macro- and microvascular architecture of soft tissue structures. Despite being currently approved for the use in hepatology and cardiology, it has remained absent from the field of spinal cord injury. The study team aims to evaluate and quantify micro- and macrovascular changes that lead to areas of hyper-perfusion as well as areas of ischemia intraoperatively in patients that undergo elective cervicothoracic posterior decompression for chronic compression. In addition, the study team aims to assess the efficacy of CEUS in detecting microvascular changes that correlate with IONM changes and predicting degree and recovery of post-operative neurologic deficits from intraoperative spinal cord injury. The study team hypothesizes that following decompression, subjects will have detectable levels of microvascular changes causing areas of hypoperfusion and reperfusion injury. Second, the study team hypothesizes that these perfusion changes will correlate with intraoperative neuromonitoring changes and can predict and prognosticate the degree of post-operative neurologic injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients consented and scheduled for posterior cervicothoracic decompression surgery with the PI for the diagnosis of cervicothoracic myeloradiculopathy
* Age 18-80

Exclusion Criteria:

* Pregnancy
* Patient's with known hypersensitivity to ultrasound contrast
* Patients with known hypersensitivity to perflutren lipid microsphere or its components, such as polyethylene glycol (PEG)
* Patients unable to actively participate in the consent process physically and/or cognitively
* Prior decompression at the intended level of decompression

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Contrast Enhanced Ultrasound to determine changes of blood flow in the spinal cord at the site of decompression. | Intra-operative (Approximately 3 hours)
  Use of Contrast Enhanced ultrasound to identify discreet areas of perfusion changes in the spinal cord of subjects that undergo spinal cord decompression.

SECONDARY OUTCOMES:
Correlation of perfusion changes measured by intra-operative Contrast Enhanced Ultrasound with neurologic outcomes measured by serial neurologic exams and functional outcomes (Frankel Grade and Modified Rankin Scale). | Clinical Monitoring (12 months)
  To assess whether discreet areas of perfusion changes seen by Contrast Enhanced ultrasound in the spinal cord intraoperatively correlate with the neurologic and functional outcomes of subjects that undergo spinal cord decompression

CONTACTS AND LOCATIONS:
Overall Officials: Brian F Saway, MD, Principal Investigator — Medical University of South Carolina; Stephen Kalhorn, MD, Principal Investigator — Medical University of South Carolina; Jessica Barley, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No